CLINICAL TRIAL: NCT05907434
Title: Cell Cycle Arrest Proteins for Early Diagnosis of Acute Kidney Injury After Solid Organ Transplant: a Prospective Observational Study
Brief Title: Cell Cycle Arrest Proteins for Early Diagnosis of Acute Kidney Injury After Solid Organ Transplant
Acronym: LUTX/OLTX_AKI
Status: Completed | Type: Observational
Sponsor: Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Giacomo Grasselli, Prof, Policlinico Hospital
Other Study IDs: 127_2022
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Acute Kidney Injury
Keywords: acute kidney injury; biomarkers; lung transplant; liver transplant
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urinary and plasma biobanking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Lung transplant recipients: Adult undergoing primary non emergent lung transplant
  Interventions: Diagnostic Test: Nephrocheck (AKI score)
- Liver transplant: Adult undergoing primary non emergent livertransplant
  Interventions: Diagnostic Test: Nephrocheck (AKI score)

INTERVENTIONS:
Diagnostic Test: Nephrocheck (AKI score) — Early biomarker of AKI
  Other Names: urinary biomarker [TIMP-2] × [IGFBP-7]

SUMMARY:
Renal failure is a common complication of lung transplant (LUTX) and orthotopic liver transplantation (OLTX). Early diagnosis of acute kidney injury (AKI) in this cohort is of utmost importance, since AKI after solid organ transplant is associated with worsened short and long-term outcomes. To now, early biomarkers of renal failure based on the measurement of cell-cycle arrest proteins have never been tested in this population.

DETAILED DESCRIPTION:
Bilateral lung transplantation (LUTX) is a surgical procedure offered to patients suffering from chronic respiratory failure. LUTX provides a survival benefit to selected patients but is associated with several short-term and long-term non-pulmonary complications.

Liver Transplantation (OLTX) is the gold-standard treatment for patients affected by end-stage liver disease or primary liver tumor. Despite its encouraging post-transplant survival, the increasing use of extended criteria donors leads to a higher incidence of post-LT complications that could affect post-LT results and quality of life.

Acute kidney failure (AKI) is frequent and associated with short-term and long-term morbidity and increased mortality. Indeed, AKI occurs in up to two-thirds of transplanted patients, with 5-13% needing renal replacement therapy (RRT), and associated with mortality ranging from 13 to 50%.

Several risk factors may favor postoperative AKI in patients undergoing solid organ transplant: preoperative (e.g., the patients' preoperative renal function and comorbidities) , intraoperative (i.e., hypoxia, hypotension, massive blood components' transfusions, use of intraoperative extracorporeal membrane oxygenation - ECMO) and postoperative (i.e., use of nephrotoxic agents as tacrolimus and antibiotics).

In patients treated with solid organ transplant, postoperative AKI increases ICU and hospital length of stay and is associated with worsened survival. At the same time, postoperative AKI is associated with an increase in end-stage renal failure and consequent chronic renal failure with potential needs of chronic RRT. Finally, AKI may determine graft dysfunction with direct and indirect mechanisms (i.e., inability to reach therapeutic targets of anti-rejection drugs).

According to the most recent guidelines (i.e., the Kidney Improving Global Outcomes (KDIGO) criteria), patients are classified as suppering postoperative AKI stage 1, stage 2, and stage 3 are diagnosed whether serum creatinine increases 1.5-1.9 times, 2-2.9 times, and >3 times from the preoperative, respectively. However, these traditional indicators of kidney function have limitations related to early and accurate identification of AKI. Furthermore, sCr has limitations in the specific context of solid organ transplant recipients, both regarding baseline patients' clinical characteristics and surgical. On the one hand, patients enlisted for transplant are usually undernourished, have reduced muscle mass, reduced protein and creatine intake, which severely limit the sensibility and sensitivity of sCr changes for AKI diagnosis. On the other hand, the need for massive fluid and blood products during sugical operation resulting in fluid overload can mask the increase in sCr, delaying the diagnosis of AKI. In addition, early detection of AKI using sCr concentrations is limited by the fact that sCr concentrations increase when renal function has already deteriorated.

Thus, novel markers capable of early and effective diagnosis of AKI in this patient population are a major clinical interest and may allow to carry out risk-mitigating clinical approaches (e.g., volume optimization, avoid nephrotoxic agents).

Cell Cycle arrest proteins have been suggested as early indicators of AKI. In particular, urinary tissue inhibitor of metalloproteinases-2 (TIMP-2) and insulin-like growth factor binding protein-7 (IGFBP-7) are biomarkers of the renal tubular cell cycle arrest at the early phase of AKI. The product of the urinary concentrations of TIMP-2 and IGFBP-7 (urinary [TIMP- 2] × [IGFBP-7]) is a promising biomarker for early prediction of AKI in various clinical settings such as out-of-hospital cardiac arrest, in critically ill patients, and following major surgery or emergency department admission .

It is possible to envision the employment of the urinary [TIMP- 2] × [IGFBP-7] index as early indicators of renal failure in patients undergoing LUTX. Thus, with this prospective observational study, the aim of the study is to test the sensitivity and specificity of this index in detecting early AKI in patients undergone LUTX and OLTX.

Hypothesis/objectives of the study:

In patients undergoing LUTX and OLTX, the urinary biomarker [TIMP-2] × [IGFBP-7] measured on the first postoperative day after LUTX was evaluated as a reliable early predictive index of postoperative AKI compared to standard KIDGO criteria.

ELIGIBILITY:
Inclusion Criteria:

* Enlistment for bilateral LUTX
* Enlistment for bilateral OLTX
* Age > 18 years
* Signed informed consent

Exclusion Criteria:

* Age < 18 years old
* Urgency enlistment
* Already undergone solid organ transplant
* Preoperative use of RRT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult undergone primary double lung transplant or liver transplantation
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
acute kidney injury | <7 days from transplant
  according to KIDGO guidelines

SECONDARY OUTCOMES:
acute kidney disease | < 90 days from transplant
  according to KIDGO guidelines

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Ca'Granda - Ospedale Maggiore Policlinico, Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Upon reasonable request